CLINICAL TRIAL: NCT04563715
Title: Regular HIV Testing and HIV Prevention Among At-Risk Latino Men in the Heartland
Brief Title: HIV Prevention Among At-risk Latinos in the Heartland
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laura R. Glasman, Associate professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32961; R01MH116787 (NIH)
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections
Keywords: HIV; Latinos; Networks; Men who have sex with men; Transgender; USA Midwest
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): HIV counseling and testing
  Interventions: Diagnostic Test: HIV counseling and testing
- Standard of Care plus Network Intervention (Experimental): Network intervention
  Interventions: Diagnostic Test: HIV counseling and testing; Behavioral: Network intervention

INTERVENTIONS:
Diagnostic Test: HIV counseling and testing — Receive HIV testing risk assessment and advice about risk reduction and future testing.
Behavioral: Network intervention — Key individuals are trained to provide advice about regular testing and risk reduction.
  Arms: Standard of Care plus Network Intervention

SUMMARY:
This study is a randomized controlled trial that evaluates the efficacy of a network intervention to promote regular HIV testing and prevention (risk reduction and PrEP awareness and referrals) among friendship networks of Latino men who have sex with men and transwomen (LMSMT) in three mid sized Midwestern cities.

DETAILED DESCRIPTION:
To benefit from early HIV diagnosis, the CDC suggests that groups at higher HIV risk get tested regularly. The study will evaluate the efficacy of an intervention to promote regular HIV testing and prevention (risk reduction and PrEP awareness and referrals) among friendship networks of Latino men who have sex with men and transwomen (LMSMT) in three midsized Midwestern cities. The intervention uses the relationships that permeate networks of LMSMT by training well-positioned members to encourage a collective response to the epidemic and to disseminate HIV testing and prevention messages and resources within the network. Thus, we will (a) recruit 36 friendship networks of LMSMT in Milwaukee, Cleveland, and Indianapolis (N ≈ 432); (b) test them for HIV and recommend that they test regularly; (c) invite key members of 18 randomly selected networks to a 4-session training to promote regular HIV testing and prevention in their networks; (d) conduct chart reviews to verify regular testing and PrEP visits and assess regular testing, PrEP visits, and risk behavior and mediators at 6, 12 and 18-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Latinx men who have sex with men or transgender women 18 or more years of age.
* Lives in the Milwaukee, Cleveland or Indianapolis area.
* Can provide informed consent.
* Additional inclusion criteria for networks: 80% or more of the network is of Latinx descent.

Exclusion Criteria:

* Cis-gender female.
* Did not have sex with men or identify as homosexual or bisexual.
* Cannot provide consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male gender at birth
Enrollment: 456 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean percentage of participants who report having tested for HIV twice in the past 12 months. | Past 12 months
  Participants will complete surveys assessing HIV testing behavior.
Mean percentage of PrEP-eligible participants who report having consulted with a provider about PrEP. | Past 6 months
  Participants will complete surveys in which they will report whether they consulted with a provider about PrEP.
Mean percentage of participants who report having had unprotected sex with a casual partner. | Past 6 months
  Participants will complete surveys in which they will report whether they had unprotected sex with a casual partner.
Mean percentage of participants who report having tested for HIV in the past 6 months. | Past 6 months
  Participants will complete surveys assessing HIV testing behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Laura R Glasman, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - Shalom Health Care Center, Indianapolis, Indiana
  - AIDS Taskforce of Greater Cleveland, Cleveland, Ohio
  - Sixteenth Street Community Health Centers, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No